CLINICAL TRIAL: NCT05792501
Title: Frequencies, Risk Factors and Outcome of Ventilation-Associated Lung Complications At Paediatric Intensive Care Unit (PICU)
Brief Title: Pulmonary Infections and Barotrauma Associated With MV IN PICU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mahmoud Ezzat, principle investigator, Assiut University
Other Study IDs: Complication Of MV IN PICU
Record Dates: First submitted 2023-01-09; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Ventilator Associated Pneumonia (VAP)
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mechanical ventilation — type of therapy that helps you breathe or breathes for you when you can't breathe on your own

SUMMARY:
This study aims to determine the incidence, risk factors and outcome of ventilation associated common complication in the PICUs at Assiut University Children Hospital in Egypt.

DETAILED DESCRIPTION:
A constellation of adverse effects and complications may be associated with mechanical ventilation,The following are the Commonest Complications of Mechanical Ventilation

1. Ventilator-associated pneumonia.
2. Ventilator-induced lung injury.
3. Ventilation induce Hemodynamic compromise leads to ARDS. Ventilator-Associated Pneumonia (VAP) It refers to nosocomial pneumonia occurring 48 hours or more after initiation of mechanical ventilation (MV)

It is the second most common HAI after blood stream infection in the paediatric age group, accounting for about 20% of all HAIs in the paediatric intensive care units (PICUs) and has a rate of 2.9- 21.6 per 1000 ventilator days.The risk factors responsible for VAP occurrence can be classified into:

A-Host related factors: include associated co-morbidities B-Device-related factors: include the endotracheal tube, the ventilation circuit, and the presence of a nasogastric or an orogastric tube.

C-Personnel related factors: include improper hand hygiene and inadequate use of personal protective equipment.

VAP is associated with increased hospital morbidity; mortality; duration of hospitalization by an average of 7-9 days per patient; and health care costs . The incidence rates of VAP are higher in developing countries with limited resources.

Ventilator-associated lung injury (VALI) It is the lung damage by application positive or negative pressure to the lung by mechanical ventilation.

The prevalence of VALI in children admitted to the paediatric intensive care unit (PICU) may approximate 10%.

Types of VALI:

* Voltrauma (This is damage caused by over-distension)
* Barotrauma (destructive entry of pressurised airway gases into the parenchyma, or into blood vessels.)
* Biotrauma (is known to upregulate pulmonary cytokine production)
* Oxygen toxicity (This is the damage caused by a high concentration of inspired oxygen)
* Recruitment /de-recruitment injury (atelectotrauma)
* Shearing injury Risk factors for VALI: blood product transfusion, acidaemia, and history of restrictive lung disease. larger tidal volume.

investigators observed lower mortality among children ventilated with Vt ~8 mL/kg actual bodyweight compared with ~10 mL/kg in a before-after retrospective study .

Ventilation induce Hemodynamic compromise leads to ARDS:

Definition: Decrease in mean arterial pressure of 60 mm Hg or an absolute decrease to a systolic blood pressure < 80 mm Hg in the first 2 hours after intubation, required treatment for LTH with vasopressors.

primary factor influencing mortality in acute respiratory distress syndrome (ARDS) Incidence: 28.6% of patients intubated in the emergency department developed post-intubation hypotension, tatistically significant association between LTH and hyper carbic (PCO2 > 50 mm) chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria:

* children aged one month to up to 16 years Intubated and connected to MV for at least 48hrs.

Exclusion Criteria:

* Neonates and cases connected to M.V less than 48 hours.

Ages: 1 Month to 16 Years | Sex: All
Age Groups: Child
Study Population: children aged one month to up to 16 years Intubated and connected to MV for at least 48hrs.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
assess right sided heart failure post ventilator acquired pneumonia | one year from april 2022 to april 2023
  use modified ross score for evaluation of heart failure post mechanical ventilation

SECONDARY OUTCOMES:
Asess the risk factors associated with barotrauma on mechanical ventilation | one year from april 2022 to april 2023
  previous chronic lung disease .previous NICU or PICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- PICU, Asyut, Assuit, Egypt

REFERENCES:
- [Background] Schouten LR, Veltkamp F, Bos AP, van Woensel JB, Serpa Neto A, Schultz MJ, Wosten-van Asperen RM. Incidence and Mortality of Acute Respiratory Distress Syndrome in Children: A Systematic Review and Meta-Analysis. Crit Care Med. 2016 Apr;44(4):819-29. doi: 10.1097/CCM.0000000000001388. PMID 26509320
- [Background] Sud S, Sud M, Friedrich JO, Wunsch H, Meade MO, Ferguson ND, Adhikari NK. High-frequency ventilation versus conventional ventilation for treatment of acute lung injury and acute respiratory distress syndrome. Cochrane Database Syst Rev. 2013 Feb 28;(2):CD004085. doi: 10.1002/14651858.CD004085.pub3. PMID 23450549